CLINICAL TRIAL: NCT04876209
Title: Reference Values of Aerobic Fitness in the Contemporary Paediatric Population: VO2max Z-scores
Brief Title: Reference Values of Aerobic Fitness in the Contemporary Paediatric Population
Acronym: SAIN&NORMES
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Department of Paediatric Cardiology and Congenital Heart Disease, German Heart Centre Munich, Germany. (Unknown); Department of Cardiology Children's Hospital, Boston, United State. (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0475
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Healthy; Obese
Keywords: Cardiopulmonary exercise test; Z score; Pediatric; VO2max; VE/VCO2 slope
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In most pediatric medical conditions, tremendous progress in pediatrics has significantly improved the overall prognosis and transferred the mortality from childhood to adulthood. Nevertheless, chronic diseases remain the leading cause of death and physical inactivity appears to be a major aggravating factor. Yet, a good physical activity has a positive impact on quality of life and prevents future health morbidities, such as obesity and cardiovascular disease. Therefore, after focusing on the survival of children with chronic diseases, more attention is being given to health-related quality of life and secondary prevention.

In this context, the cardio-pulmonary exercise test (CPET), which is a non-invasive and dynamic examination, has become the gold standard to identify subjects with impaired physical capacity and to identify the causes of their limitations (muscular, cardiac, respiratory, behavioral, etc.). Moreover, CPET is the key examination to enroll patients in personalized physical rehabilitation programs (muscle deconditioning, respiratory limitation, etc.).

Despite a growing interest in CPET and individualized rehabilitation programs for chronic diseases, the investigators still face the lack of reference values for pediatric CPET. In current practice, many CPET pediatric laboratories use the reference values of maximum oxygen uptake (VO2max) defined by Cooper et al. in 1984, from a cohort of 109 healthy children. However, their equations are linear and based on weight only. Non linear equations and the use of other anthropometric variables may be relevant in pediatrics. For instance, in the current era, normal CPET pediatric values should consider the prevalence of overweight and obesity in childhood general population (respectively 30% and 10% in Europa and 35% and 25% in North America), as well as in the population of children with chronic disease.

In the past decade, our group has developed a research program on physical capacity in children, with a focus on pediatric CPET and physical rehabilitation, from a cohort of nearly 1000 exercise tests in children. The lack of reliable pediatric reference values for VO2max, and all CPET variables as well, has become an important issue.

In this study, the investigators aim to define pediatric reference CPET values from a large cohort of 6 to 17 year-old children, using several anthropometric variables to define the most appropriate Z-scores equations (part 1). The investigators will also validate the Z-scores equations using an independent population (part 2).

DETAILED DESCRIPTION:
This cross-sectional study included healthy children from 6 to 17 years old and obese children with no other comorbidities other than those due to metabolic syndrome (hypertension, dyslipidemia, type 2 diabetes sleep apnea, hepatic steatosis). Patients refuse the use of medical data will be excluded.

Part 1 - Z-score equations: After description of the study sample, the regression method will be identified (linear, polynomial, logarithmic, spline, etc.). The main anthropometric determinants (age, gender, height, weight, BMI) will be tested, and the mathematical models that best fit to the data will be identified (use of the adjusted coefficient of determination R2). The models will calculate, for each subject, the difference between the value predicted by the model and the value actually observed (residuals of the model). The occurrence of heteroscedasticity (e.g. the circumstance in which the variability of a variable is unequal across the range of values of a second variable that predicts it) will be tested. The Z-scores will be measured by the difference between predicted values and observed values divided by the calculated standard deviation.

Part 2- Validation of Z-score equations from an independent population The validity of the Z-score equations will be tested on a cohort of 100 pediatric in 6 to 18 year-old children, from pediatric CPET laboratories that did not participate in the part 1 study. The CPET variables may be retrospectively collected from existing database or prospectively collected, but no CPET should be performed for the only purpose of the research (observational study)

ELIGIBILITY:
Part 1 - Z-score equations:

Healthy children:

Inclusion criteria

* Child from 6 to 17 years old having performed a cardio-respiratory exercise test for chest pain, dyspnea on exertion, heart murmur and whose results do not find:
* congenital heart disease (normal echocardiography and ECG)
* respiratory disease (normal FEV1 and FVC)
* Child having performed a maximal cardio-respiratory stress exercise until exhaustion.

Exclusion criteria:

* Child taking long-term drug treatment
* Child with chronic disease
* Parents' refusal to use medical data.

Obese children:

Inclusion criteria

* Child with BMI>85e percentile
* Child from 6 to 17 years old having performed a cardio-respiratory exercise test for checkup and whose results do not find:
* congenital heart disease (normal echocardiography and ECG)
* Child having performed a maximal cardio-respiratory stress exercise until exhaustion.

Exclusion criteria:

* Child taking long-term drug treatment (except for their metabolic syndrome)
* Child with chronic disease (except their metabolic syndrome)
* Parents' refusal to use medical data.

Part 2 : Validation of Z-score equations from an independent population The same criteria will be used for the patients of the Munich center and the Boston center to test our equations

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children cohort consisted of children referred to a paediatric cardiologist for a nonsevere functional symptom related to exercise (murmur, palpitation, chest pain, and dyspnoea) or for a medical sports certificate. Obese children cohort consisted of children with BMI > 85e percentile referred to a paediatric cardiologist for checkup.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
identify the parameters of an equation for calculating VO2max Z-scores | day 1
  identify the parameters of an equation for calculating VO2max Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating VO2max Z-scores | day 1
  estimate the parameters of an equation for calculating VO2max Z-scores (potentially using age, sex, height, weight or skin surface area)

SECONDARY OUTCOMES:
validity of the VO2max Z-score equations | day 1
  validity of the VO2max Z-score equations will be tested from cohort from pediatric CPET laboratories that did not participate in the part 1 study. To analyze this, we will compare the difference between the measured VO2max and the VO2max predicted by the Wassermann equation (Wassermann's predicted value - observed value) and the difference between the measured VO2max and the VO2max predicted by our equation (Gavotto's predicted value - observed value)
identify the parameters of an equation for calculating ventilatory anaerobic threshold Z-scores | 1 day
  identify the parameters of an equation for calculating ventilatory anaerobic threshold Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating ventilatory anaerobic threshold Z-scores | 1 day
  estimate the parameters of an equation for calculating ventilatory anaerobic threshold Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating VE/VCO2 slope Z-scores | 1 day
  identify the parameters of an equation for calculating VE/VCO2 slope Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating VE/VCO2 slope Z-scores | 1 day
  estimate the parameters of an equation for calculating VE/VCO2 slope Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating oxygen uptake efficiency slope Z-scores | 1 day
  identify the parameters of an equation for calculating oxygen uptake efficiency slope Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating oxygen uptake efficiency slope Z-scores | 1 day
  estimate the parameters of an equation for calculating oxygen uptake efficiency slope Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating oxygen pulse Z-scores | 1 day
  identify the parameters of an equation for calculating oxygen pulse Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating oxygen pulse Z-scores | 1 day
  estimate the parameters of an equation for calculating oxygen pulse Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating maximal respiratory frequency Z-scores | 1 day
  identify the parameters of an equation for calculating maximal respiratory frequency Z-scores (potentially using age, sex, height, weight or skin surface area)
stimate the parameters of an equation for calculating maximal respiratory frequency Z-scores | 1 day
  estimate the parameters of an equation for calculating maximal respiratory frequency Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating maximal maximal tidal volume Z-scores | 1 day
  identify the parameters of an equation for calculating maximal maximal tidal volume Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating maximal maximal tidal volume Z-scores | 1 day
  estimate the parameters of an equation for calculating maximal maximal tidal volume Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating breath reserve Z-scores | 1 day
  identify the parameters of an equation for calculating breath reserve Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating breath reserve Z-scores | 1 day
  estimate the parameters of an equation for calculating breath reserve Z-scores (potentially using age, sex, height, weight or skin surface area)
estimate the parameters of an equation for calculating maximal pet end tidal CO2 Z-scores | 1 day
  estimate the parameters of an equation for calculating maximal pet end tidal CO2 Z-scores (potentially using age, sex, height, weight or skin surface area)
identify the parameters of an equation for calculating maximal pet end tidal CO2 Z-scores | 1 day
  identify the parameters of an equation for calculating maximal pet end tidal CO2 Z-scores (potentially using age, sex, height, weight or skin surface area)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur GAVOTTO, MD, Principal Investigator — University Hospital, Montpellier; Pascal AMEDRO, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Amedro P, Matecki S, Pereira Dos Santos T, Guillaumont S, Rhodes J, Yin SM, Hager A, Hock J, De La Villeon G, Moreau J, Requirand A, Souilla L, Vincenti M, Picot MC, Huguet H, Mura T, Gavotto A. Reference Values of Cardiopulmonary Exercise Test Parameters in the Contemporary Paediatric Population. Sports Med Open. 2023 Aug 1;9(1):68. doi: 10.1186/s40798-023-00622-3. PMID 37528295
- [Background] Gavotto A, Mura T, Rhodes J, Yin SM, Hager A, Hock J, Guillaumont S, Vincenti M, De La Villeon G, Requirand A, Picot MC, Huguet H, Souilla L, Moreau J, Matecki S, Amedro P. Reference values of aerobic fitness in the contemporary paediatric population. Eur J Prev Cardiol. 2023 Jul 12;30(9):820-829. doi: 10.1093/eurjpc/zwad054. PMID 36809338